CLINICAL TRIAL: NCT02820532
Title: Influence of Couch Tracking Motion on Physiological Parameters
Brief Title: Influence of Couch Tracking Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Technical University Zurich (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-00163
Record Dates: First submitted 2016-06-20; First posted 2016-07-01 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Amplitude

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tracking (Other): The volunteers will be placed on the treatment couch. Their respiratory motion will be measured and the treatment couch will be moved accordingly. During the couch motion experiment the heartbeat, the skin humidity, the respiratory characteristics and the pupil motion will be additionally measured.
  Interventions: Device: Protura Treatment table

INTERVENTIONS:
Device: Protura Treatment table — The treatment couch will be moved according to the respiratory motion of the patient. As a reference first the respiration will be measured without couch motion, than the couch will be switched on and we will evaluate if the respiration changes due to the motion of the couch. This procedure will be repeated once.

SUMMARY:
Tumor motion increases the uncertainty in Radiation Oncology. Couch tracking can compensate for this uncertainty. However it is not known if the couch motion influences the respiratory pattern of the patients. This will be evaluated in this study on healthy volunteers.

DETAILED DESCRIPTION:
Radiation therapy is one of the main options in cancer treatments, alongside surgery and chemotherapy. Its efficacy largely depends on the absorbed radiation dose of the tumor cells. However, the irradiation of healthy cells results in negative side effects for the patient. Therefore, a big challenge in radiation therapy is to irradiate the tumor with sufficient dose, while keeping the irradiation of the healthy tissue reasonably low. Currently, the radiation treatment is planned by defining a volume enclosing the tumor, but with added margins to account for any uncertainties. These margins ensure that the tumor receives the prescribed dose.

Tumor motion contributes to the uncertainties. The tumor motions of tumors in different sites have different causes, but for this project the focus is on thoracic, liver, and adrenal gland tumors. The motion of these tumor types is mainly caused by the patient's respiration. So, the tumor motion pattern depends on the respiration pattern of the patient. The motion of lung tumors has been reported to have a peak-to-peak amplitude of up to 24 mm. Currently, the tumor motion is handled by enlarging the margins, such that the tumor is always inside the defined volume. But enlarging the margins also results in an increase of irradiated volume consisting of healthy tissue.

Tumor motion mitigation is concerned with reducing the margin increase caused by the motion of the tumor. There are several approaches to tumor motion mitigation and the one under consideration in this project is the tumor tracking approach, the technically most difficult approach. In tumor tracking the tumor motion is continuously compensated by moving the radiation source modifying the radiation beam, or moving the patient, which is denoted as couch tracking.

In couch tracking, the patient is moved by the robotic treatment couch. Such robotic treatment couches are in use with conventional, widely available C-arm linear accelerators, and, therefore, are readily available for implementing couch tracking. The patient is placed on a couch which moves in the opposite direction of the tumor motion. The goal is to minimize the patient's tumor motion relative to the radiation, which in turn allows the margins to be decreased. The margin decrease might ultimately lead to a reduction of side effects, e.g. pneumonitis.

The motion of the couch depends on the motion of the tumor, which in turn depends on the respiration of the patient. However, the couch motion may influence the patient's well being or the patient's respiration. So the question arises: Does the motion of the couch have an influence on the respiration behavior? And also: Does the motion of the couch have an influence on the well being (motion sickness)? And are the well-being and the respiration behavior connected? If the respiration behavior does depend on the couch motion, it may be necessary to control the respiration behavior. Additionally, in the study, the investigators will check an assumption in couch tracking, namely that the patient's body is rigidly fixed to the couch. If this assumption does not hold, the motion of the patient's body relative to the couch will have to be taken into account in couch tracking.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Male and Female subjects
* ≥18 and ≤100 years
* Written informed consent by the participant after information about the project
* German speaking

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Body weight exceeding 200kg

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Respiratory amplitude | baseline and 20 min
  Change of respiratory motion due to couch motion. Respiration will be measured on the chest wall using a contact-free measurement.

SECONDARY OUTCOMES:
Heart beat | baseline and 20 min
  The heart beat will be measured on the palm of the hand during the static and the couch motion phase.
Skin humidity | baseline and 20 min
  The skin humidity will be measured on the hand palm during the static and the phase in motion.
Pupil motion | baseline and 20 min
  The change in pupil motion during tracking compared to static condition will be assessed using eye tracking glasses.
Body motion | baseline and 20 min
  The influence of the couch motion on the body motion will be assessed using a surface detection system.
Motion sickness | baseline and 20 min
  With a questionaire the motion sickness is assessed, which the participants might experience during couch motion

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, MD, Principal Investigator — University Hospital Zurich, Department of Radiation Oncology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johl A, Bogowicz M, Ehrbar S, Guckenberger M, Klock S, Meboldt M, Riesterer O, Zeilinger M, Schmid Daners M, Tanadini-Lang S. Body motion during dynamic couch tracking with healthy volunteers. Phys Med Biol. 2018 Dec 19;64(1):015001. doi: 10.1088/1361-6560/aaf361. PMID 30523943
- [Derived] Johl A, Bogowicz M, Ehrbar S, Guckenberger M, Klock S, Meboldt M, Riesterer O, Zeilinger M, Schmid Daners M, Tanadini-Lang S. Unconscious physiological response of healthy volunteers to dynamic respiration-synchronized couch motion. Radiat Oncol. 2017 Nov 28;12(1):189. doi: 10.1186/s13014-017-0925-6. PMID 29183337